CLINICAL TRIAL: NCT05785728
Title: Phase 1/2, Multicenter, Open-label, First-in-human Study of DB-1202 Monotherapy in Patients With Advanced Solid Malignant Tumors to Evaluate the Tolerability, Safety, Pharmacokinetics and Antitumor Activity
Brief Title: A Study of DB-1202 Monotherapy in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DualityBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB-1202-O-1001
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor
Keywords: TGF-β; thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- DB-1202 Dose Level 1 (Experimental): Enrolled Subjects will receive a single-dose of DB-1202 at Dose Level 1 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1202
- DB-1202 Dose Level 2 (Experimental): Enrolled Subjects will receive a single-dose of DB-1202 at Dose Level 2 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1202
- DB-1202 Dose Level 3 (Experimental): Enrolled Subjects will receive a single-dose of DB-1202 at Dose Level 3 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1202
- DB-1202 Dose Level 4 (Experimental): Enrolled Subjects will receive a single-dose of DB-1202 at Dose Level 4 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1202
- DB-1202 Dose Level 5 (Experimental): Enrolled Subjects will receive a single-dose of DB-1202 at Dose Level 5 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1202
- DB-1202 Dose Level 6 (Experimental): Enrolled Subjects will receive a single-dose of DB-1202 at Dose Level 6 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1202
- DB-1202 Dose Expansion 1 (Experimental): Enrolled Subjects with locally advanced or metastatic primary thyroid cancers with pathology of epithelial tumors that originated from thyroid follicular cells will be enrolled regardless of PD-L1 expression will receive initial dose of DB-1202 Q3W under a 21-day Treatment Cycle with RP2D.
  Interventions: Drug: DB-1202
- DB-1202 Dose Expansion 2 (Experimental): Enrolled Subjects in selected solid malignant tumors can be added will receive initial dose of DB-1202 Q3W under a 21-day Treatment Cycle with RP2D.
  Interventions: Drug: DB-1202
- DB-1202 Dose Expansion 3 (Experimental): Enrolled Subjects in selected solid malignant tumors can be added will receive initial dose of DB-1202 Q3W under a 21-day Treatment Cycle with RP2D.
  Interventions: Drug: DB-1202

INTERVENTIONS:
Drug: DB-1202 — Administered I.V.

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1/2a trial to evaluate the safety and tolerability of DB-1201 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open-label, multiple-dose, FIH study. The study consists of two parts: Part 1 adopts a rule based "3 + 3" design to identify MTD/RP2D; Part 2 is a dose expansion phase to confirm the safety, tolerability and efficacy in selected solid malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old.
2. Has histologically or cytologically confirmed metastatic or locally advanced solid tumors for which no effective standard therapy existed or standard of care has failed or is not considered as an option.
3. Is capable of comprehending study procedures and risks outlined in the informed consent and is willing to provide written consent.
4. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1.
5. At least one measurable lesion as assessed by the investigator according to response evaluation criteria in solid tumors (RECIST) version 1.1 criteria.
6. Has adequate organ function within 7 days prior to initiation of the first Treatment Cycle
7. Platelet count ≥ 100 000/mm3
8. Hemoglobin (Hb) ≥ 8.5 g/dL
9. Absolute neutrophil count (ANC) ≥ 1500/mm3
10. Creatinine ≤ 1.5 × upper limit of normal (ULN), or
11. Creatinine clearance ≥ 60 mL/min (modification Cockcroft-Gault equation)

Exclusion Criteria:

1. Has a medical history of symptomatic chronic heart failure (CHF) (New York Heart Association [NYHA] classes II-IV) or serious cardiac arrhythmia requiring treatment.
2. Has a medical history of myocardial infarction or unstable angina within 6 months before Day 1.
3. Has a QTc prolongation to > 470 millisecond (ms) based on a 12-lead electrocardiogram (ECG) in triplicate.
4. Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with a history of autoimmune thyroid disease are not excluded. Subjects with vitiligo or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
5. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
6. History of primary immunodeficiency.
7. History of allogeneic organ transplant.
8. Has an uncontrolled infection requiring IV injection of antibiotics, antivirals, or antifungals.
9. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection.
10. Is a lactating mother (women who are willing to temporarily interrupt breastfeeding will also be excluded), or pregnant as confirmed by pregnancy tests performed within 7 days prior to initiation of the first Treatment Cycle.
11. Male and female subjects who are unwilling to use adequate contraceptive methods (double barrier or intrauterine contraceptive) during the study and for at least 7 months after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-28 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by CTCAE v5.0 | up to 21 days after Cycle 1 Day 1
  Percentage of participants in Part 1 with DLTs
Phase 1: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) as assessed by CTCAE v5.0 | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with AEs in Part 1 graded according to NCI CTCAE v5.0
Phase 1: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of Participants with SAEs in Part 1 graded according to NCI CTCAE v5.0
Maximum Tolerated Dose (MTD) of DB-1202 | 12 months
  MTD on the data collected during Part 1
Phase 1: Recommended Phase 2 Dose (RP2D) of DB-1202 | 12 months
  RP2D of DB-1202 based on the data collected during Part 1
Phase 2a: Percentage of Participants with Treatment Emergent adverse events (TEAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with AEs in Part 2 graded according to NCI CTCAE v5.0
Phase 2a: Percentage participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with SAEs in Part 2 graded according to NCI CTCAE v5.0
Percentage of Objective Response Rate (ORR) as assessed by RECIST 1.1. | Up to follow-up period, approximately 1 year post-treatment
  The percentage of subjects who had a best response rating of CR and PR, for Part 2 only which was maintained ≥4 weeks

SECONDARY OUTCOMES:
Phase 1 & Phase 2a: Pharmacokinetic-AUC | within 8 cycles (each cycle is 21 days)
  Area under the concentration-time curve from time 0 to infinity of DB-1202
Phase 1 & Phase 2a: Pharmacokinetic-Cmax | within 8 cycles (each cycle is 21 days)
  Maximum observed plasma concentration (Cmax) of DB-1202
Phase 1 & Phase 2a: Pharmacokinetic-Tmax | within 8 cycles (each cycle is 21 days)
  Time to Cmax of DB-1202
Phase 1 & Phase 2a: Pharmacokinetic-T1/2 | within 8 cycles (each cycle is 21 days)
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Zhao, Study Director — DualityBio Inc.
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No